CLINICAL TRIAL: NCT01719874
Title: A Phase 2a, Double-Blind, Placebo-Controlled Study TCN 032 (Human Monoclonal Antibody Directed Against the M2 Protein of Influenza A Virus) in Subjects Challenged With H3N2 Influenza A Virus
Brief Title: Influenza Virus Challenge Study to Test Monoclonal Antibody TCN-032 as a Treatment for Influenza
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Theraclone Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCN-032-002
Record Dates: First submitted 2012-10-25; First posted 2012-11-01 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Influenza
Keywords: Influenza; monoclonal antibody
MeSH Terms: conditions — Influenza, Human | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TCN-032 (Experimental): single-dose, administered intravenously
  Interventions: Biological: TCN-032
- Placebo (saline) (Placebo Comparator): single-dose, administered intravenously
  Interventions: Biological: Placebo (saline)

INTERVENTIONS:
Biological: TCN-032
  Arms: TCN-032
Biological: Placebo (saline)
  Arms: Placebo (saline)

SUMMARY:
The purpose of this study is to determine the safety and efficacy of TCN-032 given to healthy adult volunteers that have been inoculated with the influenza A virus

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years, inclusive.
* In good health with no history of major medical conditions
* Female subjects must not be pregnant or nursing
* Have not been vaccinated for influenza virus since 2006
* Serosusceptible to the challenge virus
* Non-smoker or current smoker willing/able to desist

Exclusion Criteria:

* Presence of any significant acute or chronic, uncontrolled medical or psychiatric illness
* History or evidence of autoimmune disease
* Any history during adulthood of asthma, history of COPD, pulmonary hypertension, reactive airway disease, any chronic lung condition of any etiology), or any use of a bronchodilator or other asthma medication within adulthood
* History or clinical evidence of recurrent lower respiratory tract infection
* Positive human immunodeficiency virus (HIV), hepatitis B (HBV), or hepatitis C (HCV) antibody screen
* Subject is diabetic
* History of frequent epistaxis (nose bleeds)
* Any nasal or sinus surgery within 6 months of the screening visit
* Recent and/or recurrent history of autonomic dysfunction (fainting, palpitations, etc.)
* Any laboratory test, ECG or spirometry which is abnormal and which is deemed by the Investigator(s) to be clinically significant.
* Any acute medical condition or significant past medical history of hepatic, renal, cardiovascular, pulmonary, gastrointestinal, haematological, locomotor, immunologic, ophthalmologic, metabolic, endocrine, or other diseases
* Major surgery within 3 months prior to screening visit
* Evidence of drug of abuse or positive urine Class A drug or alcohol screen prior to admission
* Subjects symptomatic with hay fever
* Subjects with a history of significant adverse reactions/allergies
* History of allergy or intolerance to oseltamivir or zanamivir.
* Health care workers (including doctors, nurses, medical students, and allied healthcare professionals) anticipated to have patient contact within 2 weeks of viral challenge.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2012-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to evaluate the effect of TCN-032 compared to placebo in the development of clinical signs and symptoms of influenza (including upper respiratory, lower respiratory, systemic and fever). | 7 days

SECONDARY OUTCOMES:
The main secondary objective is to evaluate the effect of TCN-032 compared to placebo in total virus shedding (measured by area under the curve [AUC]) from the nasal mucosa, measured by viral culture. | 7 days
Pharmacokinetics (PK) and immunogenicity of TCN-032 | up to 28 days after viral challenge
Change in haemagglutination-inhibiting antibody (HAI) titre pre-challenge to Day 28. | 28 days after viral challenge
Development of viral resistance to TCN-032 | up to 9 days after viral challenge
To evaluate the safety of subjects who undergo influenza A viral challenge, with or without treatment with TCN-032. | up to 28 days after viral challenge
The duration of influenza symptoms or pyrexia | up to 10 days
The time to peak of influenza symptoms or pyrexia | up to 10 days
The daily incidence of influenza symptoms or pyrexia. | up to 10 days
The proportion of the components of the primary objective: upper respiratory symptoms, lower respiratory symptoms, systemic influenza symptoms, pyrexia. | 7 days
The duration of the components of the primary objective: upper respiratory symptoms, lower respiratory symptoms, systemic influenza symptoms, pyrexia. | 7 days
The time to peak of the components of the primary objective: upper respiratory symptoms, lower respiratory symptoms, systemic influenza symptoms, pyrexia. | 7 days
The daily incidence of the components of the primary objective: upper respiratory symptoms, lower respiratory symptoms, systemic influenza symptoms, pyrexia. | 7 days
The proportion of any grade influenza symptoms, or pyrexia | 7 days
The duration of any grade influenza symptoms, or pyrexia | 7 days
The time to peak of any grade influenza symptoms, or pyrexia | 7 days
The daily incidence of any grade influenza symptoms, or pyrexia | 7 days
The peak value of virus shedding from the nasal mucosa measured by viral culture | up to 9 days
The time to peak of virus shedding from the nasal mucosa measured by viral culture | up to 9 days
The duration of virus shedding from the nasal mucosa measured by viral culture | up to 9 days
The daily incidence of virus shedding from the nasal mucosa measured by viral culture | up to 9 days
The AUC of virus shedding from the nasal mucosa measured by qPCR | 6 days
The peak value of virus shedding from the nasal mucosa measured by qPCR | 6 days
The time to peak of virus shedding from the nasal mucosa measured by qPCR | 6 days
The duration of virus shedding from the nasal mucosa measured by qPCR | 6 days
The daily incidence of virus shedding from the nasal mucosa measured by qPCR | 6 days
Incidence of seroconversion to viral challenge strain | up to 28 days after viral challenge
Incidence of seroprotection to viral challenge strain | up to 28 days after viral challenge
Total tissue count and total mucus weight after viral inoculation | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor L Ramos, MD, Study Director — Theraclone Sciences, Inc.
Locations (1):
- London, United Kingdom

REFERENCES:
- [Derived] Ramos EL, Mitcham JL, Koller TD, Bonavia A, Usner DW, Balaratnam G, Fredlund P, Swiderek KM. Efficacy and safety of treatment with an anti-m2e monoclonal antibody in experimental human influenza. J Infect Dis. 2015 Apr 1;211(7):1038-44. doi: 10.1093/infdis/jiu539. Epub 2014 Oct 3. PMID 25281755